CLINICAL TRIAL: NCT04433650
Title: A Person-centred Approach to Pictorial Support in Care for Children (PicPecc)
Brief Title: Pictorial Support in Person-centred Care for Children (PicPecc)
Acronym: PicPecc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Swedish Childhood Cancer Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MTI2019-0011; KP2018-0023 (Other Grant/Funding Number: SA2018-7681)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Childhood Cancer; Communication; Symptoms and Signs
Keywords: Childhood cancer; Communication; Digital application; Intervention; Pictorial support; Symptoms and Signs
MeSH Terms: conditions — Neoplasms; Communication; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: Arm 1: Treatment 1 is control and treatment 2 is intervention. Arm 2: Treatment 1 is intervention and treatment 2 is control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): The child will firstly undergo phase A without the digital reporting and communication tool.
  The child will secondly undergo phase B with the digital reporting and communication tool (i.e., A, B).
  Interventions: Device: Pictorial support in person-centred care for children (PicPecc)
- Group 2 (Experimental): The child will firstly undergo phase B with the digital reporting and communication tool.
  The child will secondly undergo phase A without the digital reporting and communication tool (i.e., B, A).
  Interventions: Device: Pictorial support in person-centred care for children (PicPecc)

INTERVENTIONS:
Device: Pictorial support in person-centred care for children (PicPecc) — Phase A: The child has the protocol for methotrexate treatment, the healthcare professionals have one workshop that containing person-centred care, universal design, distress, symptom management and the digital reporting and communication tool.
  Phase B: The child has everything in phase A. In addition, the child use the digital reporting and communication tool that has a thermometer (graded from zero (green) to ten (red)). The result of the assessment is visualized as a face (mimic and colour represents the intensity of the symptom and/or emotion (i.e., anxiety, appetite, fear/worries, how I´m feeling today, nausea, pain, sleep, and tiredness)). The digital reporting and communication tool has a body figure for location of pain, pictures for the type of pain, and an open question. There is an avatar and a gamification part, e.g., the child gets a pet after assessing the symptoms/emotions. The child reports in the app, and the child decides the frequency of assessments.

SUMMARY:
Introduction: Person-centred care is based on the assumption that every person has resources that should be used in the care situation. In order for this to happen the patient has to be able to effectively communicate his/her symptoms. This protocol describes the analysis of a digital picture-based tool for communication support for children with cancer aged 5-17 years, who undergo high-dose methotrexate treatment. The advantage of a non-linguistic based platform, beside the expected clinical outcomes, is that it can be used in multiple national studies with minimal translation.

Methods and analysis: Two studies will be conducted in a hybrid design, i.e., a crossover design will be used for the intervention (effects), and a mixed-methods design will be used for the process evaluation. Qualitative interviews will be carried out with children with cancer, their legal guardians and case-related healthcare professionals as part of the process evaluation.

The interviews will address the experiences of the intervention and frequency of use from the child's perspective. Interview transcripts will be analyzed qualitative descriptively. The digital communication tool will collect child self-reports of symptoms/emotions. The children will be monitored for biomarkers of stress and pain (neuropeptides, neurosteroids and peripheral steroids) in venous blood samples, in-app estimation levels for the children, drug consumption. Person-centeredness will be evaluated with the questionnaire Visual CARE Measure.

Ethics: Ethical approval was obtained from the Swedish Ethical Review Authority (ref 2019-02392; 2020-02601).

DETAILED DESCRIPTION:
BACKGROUND Failure in symptom relief in children with cancer leads to physical and emotional distress. Success in symptom relief is assumed to decrease distress. To initiate a person-centred approach to child-centred care means to elucidate, listen to and affirm the child´s story. Assessments of distress and symptoms are essential in symptom relief for children with cancer. However, the exclusive assessment of pain intensity can be considered a restrictive description of the experience. Novel assessment tools that give a broader description of symptoms are needed. Self-reports of symptoms are the gold standard for measuring symptoms, and strategies to achieve symptom relief to represent a dynamic and interactive process. A complex intervention has been chosen, and the project follows the Medical Research Council´s key principles and actions for consideration in the developing of the intervention.

AIM This project aims to investigate whether a person-centred communication intervention employing a new digital communication tool for children undergoing cancer treatment decrease the children's self-reported distress

Research questions:

Does adding a digital reporting and communication tool, decrease distress in children with cancer, aged 5-17 years, who undergo high-dose methotrexate treatment?

Does the adding of a digital reporting and communication tool, increase person-centredness in children with cancer, aged 5-17 years, who undergo high-dose methotrexate treatment?

Hypothesis: (i) Person-centred communication with children undergoing cancer treatment, applying a digital reporting and communication tool, will lead to reduced self-reported distress on an analogue assessment tool (paper sheet) (primary outcome), a decrease in neuropeptides, neurosteroids and peripheral steroids for stress and pain in blood, and an increased person-centeredness (secondary outcomes) (effect).

(ii) The person-centred communication is performed in child-centred ways to proactively assess children's symptoms (process) and will be evaluated with frequency of use and feasibility.

METHODS/DESIGN Study design The children will participate in a cross-over design where they are their own controls. This is a hybrid design, which evaluates both the effects and the implementation (process).

The participant is given a code in a predetermined order; the code shows whether he or she should start either with intervention (application) or with the control conditions. Randomization of the codes occurs in advance at randomizer.org, and the researcher always picks the codes in a predetermined order without knowing if it is intervention or control. This is revealed when the participant has agreed to participate in the study. Participating children participate twice, once as a control and once with e-health support Pictorial support in Person-centered care for children (PicPecc).

ELIGIBILITY:
Inclusion Criteria:

* Children with cancer, 5-17 years
* The children´s legal guardians
* Healthcare professionals who take care of these children
* The child needs to have a cognitive level of approximately five years (i.e., be able to understand a numeric rating scale (NRS)).

Exclusion Criteria:

- Children 0-4 years

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change is being assessed in self-reported distress | The self-reported distress will be collected four hours before high-dose methotrexate (T-1), when the treatment start (T0), after 24 hours (T1) and after 48 hours (T2).
  The primary outcome measure is change from baseline (T0) to 48 hours after (T2) on an 11-point NRS (0 [no distress] and 10 [worst possible distress]).

SECONDARY OUTCOMES:
Biomarkers of pain and stress in blood. | will be collected before start (T-1, T0) of the high-dose methotrexate treatment, 24 hours after start (T1), and 48 hours after start (T2).
  Levels of neuropeptides, neurosteroids and peripheral steroids.
Visual CARE Measure | This is evaluated on the VCM, which will be collected 48 hours after the start (T2) of the high-dose methotrexate treatment.
  The purpose of VCM is to give legal guardians of children <7 years old (VCM 10Q-Legal guardians), children aged 7-11 years (VCM 5Q) and adolescents aged 12 years and over (VCM 10Q) the opportunity to share their views about their experiences regarding both the meeting with the healthcare professional and their participation. If the child or the adolescent have linguistic and/or cognitive difficulties, the questionnaire for the legal guardian (10Q-Legal guardians) will be used.
Frequency of assessments of symptoms | T-1 (4 hours before treatment) - T2 (48 hours after start of treatment).
  The A phase, we will use a checklist, and in the B phase, we will record in-app. assessment levels.
Drug consumption | T-1 (4 hours before treatment) - T2 (48 hours after start of treatment).
  Drug consumption for all types of symptom relief will be recorded from the patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Nilsson, PhD, Principal Investigator — Institute of Health and Care Sciences, University of Gothenburg, Sweden; Jonas Bergquist, Professor, Study Director — Dept of Chemistry Biomedical Centre, Uppsala University, Sweden
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

REFERENCES:
- [Background] Nilsson S, Bjorkman B, Almqvist AL, Almqvist L, Bjork-Willen P, Donohue D, Enskar K, Granlund M, Huus K, Hvit S. Children's voices--Differentiating a child perspective from a child's perspective. Dev Neurorehabil. 2015 Jun;18(3):162-8. doi: 10.3109/17518423.2013.801529. Epub 2013 Aug 7. PMID 23924164
- [Background] Lin B, Gutman T, Hanson CS, Ju A, Manera K, Butow P, Cohn RJ, Dalla-Pozza L, Greenzang KA, Mack J, Wakefield CE, Craig JC, Tong A. Communication during childhood cancer: Systematic review of patient perspectives. Cancer. 2020 Feb 15;126(4):701-716. doi: 10.1002/cncr.32637. Epub 2019 Dec 10. PMID 31821552
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] O'Cathain A, Croot L, Duncan E, Rousseau N, Sworn K, Turner KM, Yardley L, Hoddinott P. Guidance on how to develop complex interventions to improve health and healthcare. BMJ Open. 2019 Aug 15;9(8):e029954. doi: 10.1136/bmjopen-2019-029954. PMID 31420394
- [Background] Nilsson S, Holstensson J, Johansson C, Thunberg G. Children's Perceptions of Pictures Intended to Measure Anxiety During Hospitalization. J Pediatr Nurs. 2019 Jan-Feb;44:63-73. doi: 10.1016/j.pedn.2018.10.015. Epub 2018 Nov 3. PMID 30683283
- [Derived] Nilsson S, Wiljen A, Bergquist J, Chaplin J, Johnson E, Karlsson K, Lindroth T, Schwarz A, Stenmarker M, Thunberg G, Esplana L, Frid E, Haglind M, Hook A, Wille J, Ohlen J. Evaluating pictorial support in person-centred care for children (PicPecc): a protocol for a crossover design study. BMJ Open. 2021 May 4;11(5):e042726. doi: 10.1136/bmjopen-2020-042726. PMID 33947726
- See also: Pictorial support in person-centred care for children — https://www.gu.se/forskning/picpecc-pictorial-support-in-person-centred-care-for-children